CLINICAL TRIAL: NCT00954707
Title: A Prospective, Randomized, Multi-Center, Double-Blind Trial to Assess the Effectiveness and Safety of Different Durations of Dual Anti-Platelet Therapy (DAPT) in Subjects Undergoing Percutaneous Coronary Intervention With the CYPHER® Sirolimus-eluting Coronary Stent (CYPHER® Stent)
Brief Title: CYPRESS - CYPHER for Evaluating Sustained Safety
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cordis US Corp. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P09-6301
Record Dates: First submitted 2009-08-06; First posted 2009-08-07 (Estimated); Results first posted 2013-10-09 (Estimated); Last update posted 2014-02-07 (Estimated); Status verified 2014-01

CONDITIONS: Coronary Artery Disease
Keywords: Atherosclerosis
MeSH Terms: conditions — Coronary Artery Disease; Atherosclerosis | interventions — Clopidogrel; Aspirin; Prasugrel Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 12m DAPT Group (Placebo Comparator)
  Interventions: Drug: Placebo & Aspirin
- 30m DAPT Group (Active Comparator)
  Interventions: Drug: Clopidogrel & Aspirin, Prasugrel & Aspirin

INTERVENTIONS:
Drug: Clopidogrel & Aspirin, Prasugrel & Aspirin — This population consists of subjects enrolled in the study who are free from death, MI, stroke, repeat coronary revascularization, major bleeding, and ST 12 months after stent implantation and who are compliant with 12 months of dual antiplatelet therapy following stent implantation and who are subsequently randomized to receive 18 months of thienopyridine treatment in addition to aspirin.
  Arms: 30m DAPT Group
Drug: Placebo & Aspirin — This population consists of subjects enrolled in the study who are free from death, MI, stroke, repeat coronary revascularization, major bleeding, and ST 12 months after stent implantation and who are compliant with 12 months of dual antiplatelet therapy following stent implantation and who are subsequently randomized to receive 18 months of placebo treatment in addition to aspirin.
  Arms: 12m DAPT Group

SUMMARY:
CYPRESS: A Prospective,Randomized,Multi-Center,Double-Blind Trial to Assess the Effectiveness and Safety of Different Durations of Dual Anti-Platelet Therapy (DAPT) in Subjects Undergoing Percutaneous Coronary Intervention with the CYPHER® Sirolimus-eluting Coronary Stent (CYPHER® Stent)

DETAILED DESCRIPTION:
During Phase I (non-randomized phase) of this study, the primary objective is to assess the rate of target lesion failure in subjects implanted with the CYPHER® stent and receiving dual antiplatelet therapy for 12 months.

During Phase II (randomized phase) of this study, the primary objective is to assess safety (major and minor bleeding), MACCE, and ST rates in subjects treated with dual antiplatelet therapy for 12 or 30 months following CYPHER® stent implantation.

*Subjects treated with the CYPHER® 2.25mm stent will be followed through 60 months.

**The last 500 patients enrolled will not be eligible for randomization.

ELIGIBILITY:
DAPT Group - Inclusion Criteria:

Phase I: Enrollment Inclusion Criteria

Subjects must meet ALL of the following inclusion criteria to be enrolled in the study:

* The subject must be 18 years of age.
* Subjects undergoing percutaneous intervention with stent deployment
* Subjects without known contraindication to dual antiplatelet therapy for at least 30 months after enrollment and stent implantation.
* The subject or Legally Authorized Representative has consented to participate and has authorized the collection and release of his/her medical information by signing the "Patient Informed Consent Form" that is approved by the Institutional Review Board or Independent Ethics Committee. The informed consent will be valid for the duration of the trial or until the subject withdraws.

DAPT Group Phase II: Randomization Inclusion Criterion at 12 months

Subjects must meet the following criterion to be eligible for randomization in the study:

* Subject is 12 Month Clear

DAPT Group - Exclusion Criteria:

Phase I: Enrollment Exclusion Criteria

Subjects will be excluded if ANY of the following exclusion criteria apply:

* Index procedure requiring use of a stent with a nominal diameter < 2.25 mm or > 3.5 mm.
* Pregnant women.
* Planned (at time of enrollment) surgery necessitating discontinuation of antiplatelet therapy within the 30 months following enrollment.
* Current medical condition with a life expectancy of less than 3 years.
* Concurrent enrollment in another device or drug study where the primary endpoint has not been reached or the device/drug might affect major endpoint outcomes in either Phase I or Phase II of the study.
* The subject may only be enrolled in the study once.
* Subjects on warfarin or similar anticoagulant therapy.
* Subjects with hypersensitivity or allergies to one of the drugs or components indicated in the Instructions for Use for the device implanted.
* Subjects unable to give informed consent.
* Subject treated with both DES and BMS during the index procedure.

DAPT Group Phase II: Randomization Exclusion Criteria at 12 months

Subjects will be excluded from randomization if any of the following criteria are met:

* Pregnant women.
* Subject switched thienopyridine type within 6 months prior to randomization
* Percutaneous coronary interventions or cardiac surgery between 6 weeks post index procedure and randomization.
* Planned surgery necessitating discontinuation of antiplatelet therapy within the 21 months following randomization.
* Current medical condition with a life expectancy of less than 3 years.
* Subjects on subsequent warfarin or similar anticoagulant therapy.
* Subjects who do not receive any CYPHER® Stent during the index procedure.

Non-DAPT Group

The following inclusion and exclusion criteria are for the Non-DAPT subjects. These criteria will be used to determine if the subject meets the near on-label definition

Non-DAPT Group - Inclusion Criteria:

Subjects must meet ALL of the following criteria to be enrolled in this study:

1. The subject must be ≥18 years of age
2. Index procedure requiring use of a stent with a nominal diameter 2.25mm to 3.5mm
3. Lesion Length ≤ 34mm
4. Up to 2 lesions in up to 2 vessels (2 in one vessel or 1 in each of 2 vessels)
5. Ejection fraction > 30%
6. Target lesion stenosis is >50% and <100% (visual estimate)
7. Female of childbearing potential must have a negative pregnancy test within 10 days prior to enrollment
8. The subject or Legally Authorized Representative has consented to participate and has authorized the collection and release of his/her medical information by signing the "Patient Informed Consent Form"

Non-DAPT Group - Exclusion criteria

And must NOT meet any of the following exclusion criteria:

1. Target Lesion includes Bifurcations with side branch diameter >2.5mm
2. Patient with excessive calcified/angulated lesion that is not suitable for stenting in the Investigator's opinion
3. Restenotic Target Lesion previously treated with a stent
4. Greater than 2 overlapping stents used to treat target lesion.
5. Target Lesion within an unprotected Left Main (LM) with ≥50% stenosis
6. Target Lesion within a coronary bypass graft (e.g., saphenous vein or arterial graft)
7. Chronic (> 3 months) Total Occlusion (CTO) Lesions, TIMI grade 0 or 1 in the target lesion
8. ST segment Elevation Myocardial Infarction (STEMI) within 30 days or non-STEMI within 72 hours
9. Renal insufficiency (creatinine >2.5 mg) or dialysis dependent
10. Lesion with visible clot
11. Patient with prior brachytherapy
12. Documented left ventricular ejection fraction is ≤30%
13. Pretreatment with devices other than conventional balloon angioplasty
14. Recipient of heart transplant
15. Subject with a life expectancy less than 1 year
16. Known allergies to the following: aspirin, all commercially available anti-platelet drugs heparin, stainless steel, contrast agent (that cannot be managed medically), or sirolimus (that cannot be managed medically);
17. Any significant medical condition which, in the Investigator's opinion, may interfere with the subject's optimal participation in the study;
18. Currently participating in an investigational drug or device study that has either not completed the primary endpoint where the prior study drug/device might affect this study's primary endpoint
19. In the Investigator's opinion, the lesion is not suitable for stenting.
20. Known bleeding or hypercoagulable disorder;
21. Known or suspected active infection at the time of the study procedures;
22. Subject is known to be pregnant
23. Subject is a prisoner, mentally incompetent, and/or alcohol or drug abuser;
24. Planned (at the time of enrollment) surgery necessitating discontinuation of anti-platelet therapy within the twelve (12) months following enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2509 (Actual)
Dates: Start 2009-08; Primary Completion 2012-01 (Actual); Study Completion 2016-03 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Simon, M.D., Principal Investigator — University Hospitals, Case Medical Center (Cleveland); David Kandzari, M.D., Principal Investigator — Piedmont Hospital, Atlanta, GA
Locations (1):
- University Hospitals, Case Medical Center (Cleveland), Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 2509 patients were enrolled from August 28, 2009 to January 14, 2011 across 139 clinical sites in the Unites States.
Pre-assignment Details: During the Phase I of this study, enrolled subjects were treated with at least one CYPHER® stent plus thienopyridine treatment and aspirin. During Phase II, approximately 1500 eligible subjects were randomized to either placebo or thienopyridine treatment. It is estimated that the Phase II results will be available for publishing by July 31, 2014.
Groups:
- All Enrolled Subjects: Subjects signed the consent forms and met all protocol defined inclusion criteria and none of the exclusion criteria.
Period: Overall Study
Arm/Group | All Enrolled Subjects
Started | 2509
Completed | 2342 (2342 Subjects completed 12-month Phase 1 follow-up; 167 subjects didn't complete the Phase 1.)
Not Completed | 167
Not completed — Death | 34
Not completed — Withdrawal by Subject | 100
Not completed — Lost to Follow-up | 33

BASELINE CHARACTERISTICS:
Population: Enrolled subjects were those who signed the informed consent and had met all of the inclusion and none of the exclusion criteria, and the target lesion had been successfully crossed with the intracoronary guidewire which was positioned intraluminally in the distal vessel. Enrolled subjects were also Intent to Treat (ITT).
Groups:
- CYPHER® Stent: The CYPHER® Sirolimus-eluting Coronary Stent is a BX Velocity stent design and is laser cut from 316L stainless steel seamless tubing and electropolished. The stent design is intended to balance radial strength and "closed cell" architecture with longitudinal flexibility in both unexpanded and expanded forms. The design can be broken into two distinct components: the radial expansion ring segments and the flexible connectors in an alternating fashion.
Arm/Group | CYPHER® Stent
Number analyzed (Participants) | 2509
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1368
  >=65 years | 1141
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.26 (10.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 785
  Male | 1724
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 132
  Not Hispanic or Latino | 2293
  Unknown or Not Reported | 84
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 6
  Asian | 37
  Native Hawaiian or Other Pacific Islander | 6
  Black or African American | 185
  White | 2225
  More than one race | 0
  Unknown or Not Reported | 50
Region of Enrollment [Number; unit: participants]
  United States | 2509

OUTCOME MEASURES:

1. Primary Outcome: Phase I: the Rate of Target Lesion Failure (TLF)
Description: Target lesion failure (TLF) is defined as clinically-driven target lesion revascularization, target vessel myocardial infarction, or cardiac death that could not be clearly attributed to a vessel other than the target vessel at 12 months.
Time Frame: 12 months
Population: Active subjects in the ITT population at 12-month post procedure
Measure: Number; unit: participants
Arm/Group | CYPHER® Stent
Number analyzed (Participants) | 2322
participants | 149
Statistical Analysis 1: Comparison: CYPHER® Stent; Test type: Superiority or Other; Rate of TLF at 12-month (%) = 6.4, 95% CI 2-sided [5.5 to 7.5]

2. Secondary Outcome: Rate of Device Success
Description: A study device success is defined as achievement of a final residual diameter stenosis of < 50% (by QCA), using the assigned device only. If QCA is not available, the visual estimate of diameter stenosis is used.
Time Frame: From post- procedure to hospital discharge, up to 39 days
Population: The total number of devices the Intent-to-Treat patients used in the study.
Measure: Number; unit: Devices
Units Other Than Participants: Devices
Arm/Group | CYPHER® Stent
Number analyzed (Participants) | 2509
Number analyzed (Devices) | 3271
Devices | 3205
Statistical Analysis 1: Comparison: CYPHER® Stent; Test type: Superiority or Other; Rate of device success (%) = 98.0, 95% CI 2-sided [97.4 to 98.4]

3. Secondary Outcome: Rate of Lesion Success
Description: Lesion success is defined as the attainment of < 50% residual stenosis (by Quantitative coronary angiography (QCA)) using any percutaneous method.
Time Frame: From post- procedure to hospital discharge, up to 39 days
Population: The total number of lesions the Intent-to-Treat population had at the beginning of the study
Measure: Number; unit: Lesions
Units Other Than Participants: Lesions
Arm/Group | CYPHER® Stent
Number analyzed (Participants) | 2509
Number analyzed (Lesions) | 3271
Lesions | 3264
Statistical Analysis 1: Comparison: CYPHER® Stent; Test type: Superiority or Other; Rate of lesion success (%) = 99.8, 95% CI 2-sided [99.6 to 99.9]

4. Secondary Outcome: Rate of Procedure Success
Description: Procedure success is defined as the achievement of a final diameter stenosis of < 50% (by QCA) using any percutaneous method, without the occurrence of death, Myocardial infarction (MI), or repeat coronary revascularization of the target lesion during the hospital stay.
Time Frame: From post- procedure to hospital discharge, up to 39 days
Population: Intent-to-Treat Population
Measure: Number; unit: participants
Arm/Group | CYPHER® Stent
Number analyzed (Participants) | 2509
participants | 2444
Statistical Analysis 1: Comparison: CYPHER® Stent; Test type: Superiority or Other; Rate of procedure success (%) = 97.7, 95% CI 2-sided [97.0 to 98.2]

5. Secondary Outcome: Rate of Clinically-driven Target Lesion Revascularization (TVR)
Description: Defined as any "clinically-driven" repeat percutaneous intervention of the target lesion or bypass surgery of the target vessel. Clinically-driven revascularizations are those in which the subject has a positive functional study, ischemic ECG changes at rest in a distribution consistent with the target vessel, or ischemic symptoms, and an in-lesion diameter stenosis ≥50% by QCA.
Time Frame: 12 Months
Population: ITT Population patients with the specific event prior to end of follow-up plus patients without that event but with death or adequate follow-up (within 1 month prior to end of scheduled 12 months follow-up)
Measure: Number; unit: participants
Arm/Group | CYPHER® Stent
Number analyzed (Participants) | 2318
participants | 98
Statistical Analysis 1: Comparison: CYPHER® Stent; Test type: Superiority or Other; Rate of Clinically-driven TLR (%) = 4.2, 95% CI 2-sided [3.45 to 5.13]

6. Secondary Outcome: Rate of Clinically Driven Target Vessel Revascularization (TVR)
Description: Defined as any clinically driven repeat percutaneous intervention of the target vessel or bypass surgery of the target vessel. Clinically-driven revascularizations are those in which the subject has a positive functional study, ischemic ECG changes at rest in a distribution consistent with the target vessel, or ischemic symptoms, and an in-lesion diameter stenosis ≥50% by QCA.
Time Frame: 12 months
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | CYPHER® Stent
Number analyzed (Participants) | 2318
participants | 124
Statistical Analysis 1: Comparison: CYPHER® Stent; Test type: Superiority or Other; Rate of Clinically-driven TVR (%) = 5.8, 95% CI 2-sided [4.87 to 6.81]

7. Secondary Outcome: Rate of Target Vessel Failure (TVF)
Description: Defined as target vessel revascularization, recurrent infarction, or cardiac death that could not be clearly attributed to a vessel other than the target vessel.
Time Frame: 12 Months
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | CYPHER® Stent
Number analyzed (Participants) | 2323
participants | 184
Statistical Analysis 1: Comparison: CYPHER® Stent; Test type: Superiority or Other; Rate of Target vessel failure (%) = 7.92, 95% CI 2-sided [6.85 to 9.09]

8. Secondary Outcome: Rate of Major Adverse Cardiac Events (MACE)
Description: MACE includes Death, myocardial infarction, emergent bypass surgery, or target lesion revascularization at 12 months
Time Frame: 12 Months
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | CYPHER® Stent
Number analyzed (Participants) | 2322
participants | 172
Statistical Analysis 1: Comparison: CYPHER® Stent; Test type: Superiority or Other; Rate of MACE (%) = 7.41, 95% CI 2-sided [6.37 to 8.55]

9. Secondary Outcome: Rate of Protocol Defined Stent Thrombosis (ST)
Description: Protocol defined ST includes early and late ST. Early thrombosis is defined as composite thirty-day ischemic endpoint including death, Q-wave myocardial infarction, or subabrupt closure requiring revascularization. Late thrombosis is defined as myocardial infarction occurring > 30 days after the index procedure and attributable to the target vessel with angiographic documentation (site reported or by qualitative coronary angiography) of thrombus or total occlusion at the target site and freedom from an interim revascularization of the target vessel.
Time Frame: 12 Months
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | CYPHER® Stent
Number analyzed (Participants) | 2313
participants | 21
Statistical Analysis 1: Comparison: CYPHER® Stent; Test type: Superiority or Other; Rate of protocol defined ST (%) = 0.91, 95% CI 2-sided [0.56 to 1.38]

10. Secondary Outcome: Rate of Academic Research Consortium (ARC) Defined Stent Thrombosis (ST)
Description: ARC defined ST classifies ST by type - definite, probable, possible; by timing - acute, sub-acute, late, very late. Definite includes angiographic or pathologic confirmation; probable includes Any unexplained death within the first 30 days or Any MI (related to documented acute ischemia and without another obvious cause) in the territory of the stent; Possible includes Any unexplained death > 30 days. Acute includes those ≤ 24 hours post procedure; sub-acute includes those > 24 hours to ≤ 30 days post procedure; and late includes those > 30 days to ≤ 1 year post procedure; and very late includes those > 1 year post procedure.
Time Frame: 12 Months
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | CYPHER® Stent
Number analyzed (Participants) | 2313
participants | 26
Statistical Analysis 1: Comparison: CYPHER® Stent; Test type: Superiority or Other; Rate of ARC defined ST (%) = 1.12, 95% CI 2-sided [0.74 to 1.64]

11. Secondary Outcome: Rate of Protocol Defined Major Bleeding Complications
Description: Defined by the Global Use of Strategies to Open Occluded Coronary Arteries (GUSTO) classification, including severe and moderate bleeding combined.
Time Frame: 12 Months
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | CYPHER® Stent
Number analyzed (Participants) | 2314
participants | 71
Statistical Analysis 1: Comparison: CYPHER® Stent; Test type: Superiority or Other; Rate of major bleeding complications (%) = 3.07, 95% CI 2-sided [2.40 to 3.85]

12. Secondary Outcome: Rate of Cardiac Death
Description: Include all deaths due to cardiac causes.
Time Frame: 12 Months
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | CYPHER® Stent
Number analyzed (Participants) | 2313
participants | 18
Statistical Analysis 1: Comparison: CYPHER® Stent; Test type: Superiority or Other; Rate of cardiac death (%) = 0.78, 95% CI 2-sided [0.46 to 1.23]

13. Secondary Outcome: Rate of Non-cardiac Death
Description: Include all deaths due to non-cardiac causes.
Time Frame: 12 Months
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | CYPHER® Stent
Number analyzed (Participants) | 2313
participants | 16
Statistical Analysis 1: Comparison: CYPHER® Stent; Test type: Superiority or Other; Rate of non-cardiac death (%) = 0.69, 95% CI 2-sided [0.40 to 1.12]

ADVERSE EVENTS:
Arm/Group | CYPHER® Stent
Serious Adverse Events (participants affected / at risk) | 34/2509
Other Adverse Events (participants affected / at risk) | 414/2509
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CYPHER® Stent (N=2509)
Cardiac Death (Cardiac disorders) | 18 (18)
Non-cardiac death (General disorders) | 16 (16)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CYPHER® Stent (N=2509)
Angina pectoris (Cardiac disorders) | 108 (150)
Angina unstable (Cardiac disorders) | 53 (77)
Coronary artery disease (Cardiac disorders) | 43 (64)
Coronary artery occlusion (Cardiac disorders) | 31 (34)
Myocardial infarction (Cardiac disorders) | 76 (99)
Catheter site haematoma (General disorders) | 39 (40)
In-stent coronary artery restenosis (Injury, poisoning and procedural complications) | 28 (46)
Cardiac enzymes increased (Investigations) | 26 (28)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 27 (30)
Coronary artery dissection (Cardiac disorders) | 79 (80)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days